CLINICAL TRIAL: NCT01269866
Title: Duloxetine (Cymbalta) in the Reduction of Pain Severity in Patient With Systemic Lupus Erythematosus: A Pilot Study
Brief Title: Study of Duloxetine in the Reduction of Pain in Patient With Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Jesus Gutierrez Stone (Other)
Responsible Party: Sponsor-Investigator, Dr. Jesus Gutierrez Stone, MD, Brain Resource Center
Organization: Brain Resource Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F1J-US-X059
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus Pain; Lupus; Pain; Systemic Lupus Erythematosus; Duloxetine; Cymbalta
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cymbalta (Other): Cymbalta 60 to 120 mg
  Interventions: Drug: Cymbalta

INTERVENTIONS:
Drug: Cymbalta — Cymbalta 60 to 120 mg PO QD
  Other Names: Duloxetine

SUMMARY:
The purpose of this study is to determine whether Duloxetine (cymbalta) can reduce pain severity in patient with Systemic Lupus Erythematosus.

DETAILED DESCRIPTION:
Duloxetine (Cymbalta) is a reuptake inhibitor of both serotonin and norepinephrine. By increasing levels of serotonin and norepinephrine, the descending inhibitory pain pathways may function better. These pathways lessen the perception of pain. Results of double blind, placebo controlled, clinical trials investigating the effectiveness of Duloxetine (Cymbalta) have shown that at doses of 60 mg once a day or 60 mg twice a day, Duloxetine (Cymbalta) demonstrated significantly higher rates of treatment response for pain when compared to placebo.

Given the positive findings in other clinical trial studies for Duloxetine (Cymbalta) such as Diabetic Peripheral Neuropathy (Raskin et al., 2005) and Fibromyalgia (e.g. Arnold et al., 2005), the investigators hypothesize that Duloxetine (Cymbalta) may reduce the pain severity, frequency and intensity of exacerbations in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Systemic Lupus Erythematosus (SLE) according to the American College of Rheumatology (ACR) classification criteria, before visit 1.
2. Able to swallow all required medication without opening or crushing.
3. Male or female outpatient 18-65 years old at visit 1.
4. Painful physical symptoms with a frequency > or equal to 2 times per week.
5. Painful physical symptoms with a score > or equal to 4 on the BPI- SF average pain question at visits 1 and 2.
6. Clinical Global Impression of Severity (CGI-S) score 3 or higher at visit 1.
7. Able to speak, read and provide informed consent.
8. Judged by the investigator to be reliable and agree to keep all appointments.

Exclusion Criteria:

1. Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit.
2. Pregnancy, nursing. Women of child-bearing potential (not surgically sterilized and between menarche and 1 year postmenopausal) who are not using a medically accepted means of contraception (For example, oral contraceptive, contraceptive patch, implant, Depo-Provera®, Norplant®, reliable barrier method/devices [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices]
3. Positive urine drug screen for any substance of abuse. Note: If the subject has a positive drug screen for a substance at Visit 1, a retest may be performed prior to Visit 2 if, in the judgment of the investigator, there is an acceptable explanation for the positive result. A retest is not required for a positive result for benzodiazepines or hypnotics if the investigator confirms use is within protocol criteria.
4. Serious medical illness, including any cardiovascular, hepatic, renal respiratory hematologic, endocrinologic or neurologic disease, or significant laboratory abnormality as judged by investigator.
5. Substance/alcohol abuse or dependency in the last 6 months.
6. History of serious suicide attempt or subject judged clinically to be at serious suicidal risk in the opinion of the investigator.
7. Uncontrolled narrow angle glaucoma.
8. Known hypersensitivity to Duloxetine or any active ingredients.
9. Treatment with a MAOI within 14 days prior to Visit 2 or have the potential need to use an MAOI during the study or within 5 days of discontinuation of study drug. (See Concomitant Medication List)
10. Have epilepsy or history of seizure disorder.
11. Use of any of the prohibited medications including thioridazine (Mellaril), or all the potent CYP1A2 inhibitors, that use of these drugs are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in the Brief Pan Inventory average pain questionnaire | Up to 8 weeks
  This is a pilot study designed to explore the efficacy of Duloxetine (Cymbalta) 60 mg to 120 mg once daily (QD) on the reduction of pain in patients with Lupus pain. The primary objective will be measured by comparing changes from baseline and end of study in:
  1. The Brief Pain Inventory (BPI-SF) average pain questionnaire.

SECONDARY OUTCOMES:
1. Change in Patient Global Impression of Improvement (PGI-I) score 2. Change in Montgomery Asberg Depression Rating Scale (MADRS) Total Score. 3. Change in Clinician Global of Impression (CGI) score | Up to 8 weeks
  1. Change in Patient Global Impression of Improvement (PGI-I) score
  2. Change in Montgomery Asberg Depression Rating Scale (MADRS) Total Score.
  3. Change in Clinician Global of Impression (CGI) score

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Gutierrez Stone, MD, Principal Investigator — Brain Resouce Center
Locations (1):
- Brain Resource Center, New York, New York, United States

REFERENCES:
- See also: Click here for more information about this study — http://brainresourcecenter.com